CLINICAL TRIAL: NCT00132002
Title: Phase II Study of Suberoylanilide Hydroxamic Acid (SAHA) (NSC 701852) as Salvage Therapy in Metastatic Breast Cancer
Brief Title: Suberoylanilide Hydroxamic Acid in Treating Patients With Progressive Stage IV Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Early termination for discouraging results
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02836; PHII-62; N01CM62209 (NIH); CDR0000438776 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2005-08-16; First posted 2005-08-19 (Estimated); Results first posted 2015-03-19 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2013-02

CONDITIONS: Male Breast Cancer; Recurrent Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms | interventions — Vorinostat

ARMS (1):
- Treatment (vorinostat) (Experimental): Patients receive oral suberoylanilide hydroxamic acid twice daily on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: vorinostat; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: vorinostat — Given PO
  Other Names: L-001079038; SAHA; suberoylanilide hydroxamic acid; Zolinza
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well suberoylanilide hydroxamic acid works in treating patients with progressive stage IV breast cancer. Drugs used in chemotherapy, such as suberoylanilide hydroxamic acid, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Suberoylanilide hydroxamic acid may also stop the growth of tumor cells by blocking some of the enzymes needed for cell growth

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the response rate in patients receiving SAHA for stage IV breast cancer.

SECONDARY OBJECTIVES:

I. Time to progression. II. Overall survival. III. Toxicity profile. IV. Assessment of potential biological correlates.

OUTLINE: This is a multicenter study.

Patients receive oral suberoylanilide hydroxamic acid twice daily on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed stage IV adenocarcinoma of the breast; tumor blocks and/or slides from original diagnosis or metastatic work-up must be available for correlative studies
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as > 20 mm with conventional techniques or as > 10 mm with spiral CT scan
* Prior adjuvant therapy, and up to 2 lines of prior chemotherapy (including trastuzumab containing regimens in Her-2 positive patients) for metastatic disease are allowed; prior radiation therapy is allowed, prior hormonal therapy is allowed
* Life expectancy of greater than 6 months
* Performance status: ECOG 0- 2
* Absolute neutrophil count >= 1,000/μl
* Platelets >= 100,000/μl
* Serum creatinine =< 1.6 mg/dl or calculated measured clearance >= 60 cc/min
* Total bilirubin =< 2 mg/dL
* AST and ALT =< 3 times institutional upper normal level
* Eligibility of patients receiving any medications or substances known to affect or with the potential to affect the activity or pharmacokinetics of SAHA will be determined following review by the Principal Investigator
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document
* Patients should not have taken valproic acid for at least two weeks prior to study entry

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients may not be receiving any other investigational agents
* Patients with known brain metastases are excluded from this clinical trial unless the metastases are controlled after therapy and have not been treated with steroids within the past two months
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to SAHA; these compounds include sodium butyrate, trichostatin A (TSA), trapoxin (TPX), MS-27-275 and depsipeptide
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because SAHA is a HDAC inhibitor agent with an unknown potential for teratogenesis; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with SAHA, breastfeeding should be discontinued if the mother is treated with SAHA
* HIV-positive patients receiving combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with SAHA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2005-06; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thehang Luu, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope, Duarte, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Vorinostat, 200 mg orally twice daily, was administered for the first 14 days of each 21 day cycle. Treatment was continued unless either disease progression was determined, the patient requested to be withdrawn from the study, or excessive toxicity was noted.
Period: Overall Study
Arm/Group | Arm 1
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1
Number analyzed (Participants) | 14
Age, Continuous [Median (Full Range); unit: years] | 60 [37 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Objective Tumor Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Up to 8 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1
Number analyzed (Participants) | 14
percentage of participants | 0

2. Secondary Outcome: Overall Survival
Description: Estimated using the product-limit method of Kaplan and Meier.
Time Frame: From the initial date of treatment to time of death, up to 5 years.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm 1
Number analyzed (Participants) | 14
Months | 24 [17.4 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.

3. Secondary Outcome: Progression-free Survival
Description: Estimated using the product-limit method of Kaplan and Meier. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: From start of treatment to the time of documented progression, assessed up to 5 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm 1
Number analyzed (Participants) | 14
Months | 2.6 [1.4 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.

ADVERSE EVENTS:
Time Frame: Adverse events occured over a period of 1 year and 7 months.
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Arm/Group | Arm 1
Serious Adverse Events (participants affected / at risk) | 3/14
Other Adverse Events (participants affected / at risk) | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=14)
Disease progression (General disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=14)
Hemoglobin decreased (Blood and lymphatic system disorders) | 9 (20)
Constipation (Gastrointestinal disorders) | 4 (9)
Diarrhea (Gastrointestinal disorders) | 6 (12)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 2 (3)
Mucositis oral (Gastrointestinal disorders) | 3 (5)
Nausea (Gastrointestinal disorders) | 12 (32)
Vomiting (Gastrointestinal disorders) | 7 (7)
Edema limbs (General disorders) | 2 (2)
Fatigue (General disorders) | 11 (29)
Pain (General disorders) | 3 (3)
Alanine aminotransferase increased (Investigations) | 4 (6)
Alkaline phosphatase increased (Investigations) | 6 (10)
Aspartate aminotransferase increased (Investigations) | 12 (38)
Creatinine increased (Investigations) | 3 (5)
Hyperbilirubinemia (Investigations) | 2 (2)
Leukopenia (Investigations) | 6 (15)
Lymphopenia (Investigations) | 10 (26)
Platelet count decreased (Investigations) | 6 (11)
Weight loss (Investigations) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 3 (3)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 8 (13)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 9 (22)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (8)
Hypokalemia (Metabolism and nutrition disorders) | 4 (5)
Hyponatremia (Metabolism and nutrition disorders) | 4 (6)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (3)
Serum phosphate decreased (Metabolism and nutrition disorders) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (8)
Joint pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (4)
Speech disorder (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (3)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (3)
Bladder pain (Renal and urinary disorders) | 1 (2)
Proteinuria (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (6)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 (2)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was terminated early after the first stage of a two-stage design, allowing for early termination for discouraging results

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less